CLINICAL TRIAL: NCT02567240
Title: A Novel Approach to Harvest Islets for Autologous Islet Transplantation
Brief Title: Carbon Monoxide-Saturated Medium for Islet Isolation
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Medical University of South Carolina (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Other
Other Study IDs: Pro00040035
Record Dates: First submitted 2015-10-01; First posted 2015-10-02 (Estimated); Last update posted 2019-01-04 (Actual); Status verified 2019-01

CONDITIONS: Chronic Pancreatitis
MeSH Terms: conditions — Pancreatitis, Chronic

STUDY DESIGN:
Who Masked: Participant, Care Provider
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Carbon monoxide-bubbled mediums (Experimental): Islets will be harvested with Carbon monoxide-saturated mediums
  Interventions: Other: Carbon monoxide-bubbled mediums
- Normal mediums (No Intervention): Islets will be harvested with regular mediums

INTERVENTIONS:
Other: Carbon monoxide-bubbled mediums — Islets will be harvested with carbon monoxide bubbled mediums
  Arms: Carbon monoxide-bubbled mediums

SUMMARY:
The goal of this study is to determine whether harvesting islets using carbon monoxide (CO)-saturated mediums can protect islet cell from death after autologous islet transplantation in patients with chronic pancreatitis.

DETAILED DESCRIPTION:
Investigators plan to harvest human islets using carbon monoxide-saturated mediums. Survival and function of transplanted islets will be compared with islets harvested using regular mediums.

ELIGIBILITY:
Inclusion Criteria:

1. Chronic pancreatitis patient selected for total pancreatectomy and islet autotransplantation.
2. Age between 18-69.

Exclusion Criteria:

1. Had prior pancreatic surgeries.

Note: The study was initially designed only to enroll diabetes free patients. To increase enrollment, we extended the inclusion criteria by allowing patients who are pre-diabetic to participate the study. This revision was approved by the MUSC IRB on 11/10/2015.

Ages: 18 Years to 69 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 16 (Actual)
Dates: Start 2015-01; Primary Completion 2018-10 (Actual); Study Completion 2018-12 (Actual)

PRIMARY OUTCOMES:
Area under the curve during mixed meal tolerance test | 6 months

CONTACTS AND LOCATIONS:
Overall Officials: Hongjun Wang, Ph.D, Principal Investigator — Medical University of South Carolina
Locations (1):
- GI Surgery, Medical University of South Carolina, Charleston, South Carolina, United States